CLINICAL TRIAL: NCT05070533
Title: Interventions to Prevent Falls in Elderly People Who Live at Home. PRECAISAL Study
Brief Title: Interventions to Prevent Falls. PRECAISAL Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of Covid19
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRS 1985/B/19
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Accidental Falls; Old Age; Debility; Activity, Motor
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual treatment (Active Comparator): The strength and balance activities of the LiFE program will be carried out. Participants will receive 7 home visits and will be given the support material for the manual (diptychs, pictures, etc.).
  Interventions: Behavioral: Individual treatment
- Groupal treatment (Experimental): The strength and balance activities of the LiFE program will be carried out. Participants will be invited to participate in groups of about 8 - 12 people in community venues.
  Interventions: Behavioral: Groupal treatment

INTERVENTIONS:
Behavioral: Individual treatment — Participants will receive 7 home visits to implement the program.
  Arms: Individual treatment
Behavioral: Groupal treatment — Subjects will participate in groups of about 8 - 12 to implement the program.
  Arms: Groupal treatment

SUMMARY:
This study aims to guide older people living in the community on appropriate strategies within a fall prevention program. This program is aimed at training in physical exercises carried out through group workshops or at preventing risk situations at home.

DETAILED DESCRIPTION:
Two-arm, non-blind, non-inferiority experimental design. Multicenter, randomized trial.

The study tries to assess whether a group intervention following the principles of the LiFE program is no less effective than individual intervention in reducing the incidence of falls.

ELIGIBILITY:
Inclusion Criteria:

* Older than 70 years
* Live at your address
* Are at risk of falls
* Timed Up and Go Test time timed ≥ 12 seconds
* Able to walk 200 meters without personal assistance
* Speak and read in Spanish

Exclusion Criteria:

* Perform moderate to vigorous physical activity> 150 min / week in the last 3 months
* Present any of the following medical conditions:

  * Heart failure (New York Heart Association class III and IV)
  * Recent stroke (<6 months)
  * Parkinson's disease
  * In active cancer treatment (last 6 months)
  * Class III and IV chronic obstructive pulmonary disease
  * Unstable fracture of the lower limb
  * Lower limb amputated
  * Treatment for less than 6 months of depression
  * Uncontrolled resting blood pressure of a systolic pressure> 160 or a diastolic pressure> 100 or more
  * Not being available for home visits within 11 weeks of the initial assessment: having planned trips or transfers of more than 2 months within the first 6 months of the study
  * Moderate to severe cognitive impairment (Mini Mental cognitive assessment <23)
  * Current participation in another scientific intervention trial.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of falls | 6 months
  Number of falls in relation to the degree of physical activity
Physical activity | 9 days
  It will be evaluated with a digital pedometer
Cost-effectiveness | 6 months
  Evaluated by the incremental cost-effectiveness ratio
Health effects | 6 months
  They are measured using quality-adjusted life years (QALYs) based on the EQ-5D-5

SECONDARY OUTCOMES:
Fear of falling | 6 months
  It will be assessed using the Short Falls International Scale of Efficacy. This scale measures of "concerns about falling". This scale has 7 items with a Likert scale with 4 options: 1) not at all concerned, 2) somewhat concerned, 3) fairly concerned, and 4) very concerned.
Adherence to exercise | 6 months
  It will be assessed using the Exercise Adherence Rating Scale (EARS). This scale is composed of 16 items and they were scored using a 5-point Likert scale (0 = completely agree to 4 = completely disagree) with a possible summed score range from 0 to 64.

CONTACTS AND LOCATIONS:
Overall Officials: Luis García-Ortiz, Study Chair — Primary Health Care Research Unit
Locations (1):
- Infosalud, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No